CLINICAL TRIAL: NCT07068165
Title: A Randomized Controlled Study of the Efficacy and Safety of Lenalidomide in the Treatment of Active IgG4-RD
Brief Title: A Randomized Controlled Study of the Efficacy and Safety of Lenalidomide in the Treatment of Active IgG4-related Disease
Acronym: IgG4-RD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Vice director of rheumatology department, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-25PJ0175
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-04

CONDITIONS: IgG4 Related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 5mg lenalidomide group (Experimental): Lenalidomide 5mg/d combined with prednisone, prednisone at an initial dose of 0.6-0.8mg/kg/d for 2-4 weeks, then reduced by 5mg every 1-2 weeks until discontinued (within 24 weeks)
  Interventions: Drug: 5mg lenalidomide
- 10 mg lenalidomide group (Experimental): Lenalidomide 10mg/ day combined with prednisone, the initial dose of prednisone was 0.6-0.8mg/kg/ day for 2-4 weeks, then 5mg every 1-2 weeks until withdrawal (within 24 weeks).
  Interventions: Drug: 10mg lenalidomide
- Prednisone monotherapy group (Active Comparator): The initial dose of prednisone was 0.6-0.8mg/kg/ day for 2-4 weeks, followed by 5mg every 1-2 weeks until withdrawal (within 24 weeks).
  Interventions: Drug: Prednisone monotherapy

INTERVENTIONS:
Drug: 5mg lenalidomide — Lenalidomide 5mg/d combined with prednisone, prednisone at an initial dose of 0.6-0.8mg/kg/d for 2-4 weeks, then reduced by 5mg every 1-2 weeks until discontinued (within 24 weeks)
  Arms: 5mg lenalidomide group
Drug: 10mg lenalidomide — Lenalidomide 10mg/ day combined with prednisone, prednisone at an initial dose of 0.6-0.8mg/kg/ day for 2-4 weeks, then reduced by 5mg every 1-2 weeks until discontinued (within 24 weeks)
  Arms: 10 mg lenalidomide group
Drug: Prednisone monotherapy — The initial dose of prednisone was 0.6-0.8mg/kg/ day for 2-4 weeks, followed by 5mg every 1-2 weeks until withdrawal (within 24 weeks).
  Arms: Prednisone monotherapy group

SUMMARY:
For patients with active proliferative IgG4-RD, we plan to conduct a 52-week prospective randomized controlled trial to compare the efficacy and safety of 5mg lenalidomide plus prednisone, 10mg lenalidomide plus prednisone, and prednisone alone, so as to find new treatment measures for patients with proliferative IgG4-RD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 75 years who meet the 2019 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification criteria for IgG4-RD；
2. Patients with active disease: For patients with initial treatment or relapse after drug withdrawal, active disease is defined as having an IgG4-RD Response Index (RI) of at least 2 points in at least one organ at the time of screening; for those experiencing relapse while on treatment, active disease is defined as having an IgG4-RD RI of at least 3 points in at least one organ at the time of screening；
3. Patients with the clinical subtype of proliferative IgG4-RD；
4. Patients who have no plans for pregnancy within the next 18 months and who agree to use reliable contraceptive measures during the study period；

Exclusion Criteria:

1. IgG4-RD patients with only fibrotic features;
2. Absolute neutrophil count <1.5×10^9 /L or platelet count <100×10^9/L;
3. Creatinine clearance less than 60 ml/ min;
4. Liver function Child-Pugh grade B or above;
5. Chronic active infection requiring systemic treatment;
6. Diagnosed with malignant tumor in the past five years;
7. Patients with a history of thrombosis;
8. Using biological agents within six months;
9. Known to be allergic to lenalidomide or thalidomide;
10. Pregnant or lactating women;
11. Patients with any other medical conditions or for specific reasons judged by the investigator to be ineligible to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2028-07-20 (Estimated); Study Completion 2028-08-20 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate at 52 weeks | "From enrollment to the end of treatment at 52 weeks

SECONDARY OUTCOMES:
Treatment response rate | At 4, 12, 24, 36, 52 weeks
IgG4 - RD RI change | At 4, 12, 24, 36, 52 weeks
Change of IgG4-RD damage index (DI) | At 4, 12, 24, 36, 52 weeks
physician's overall assessment of disease activity | At 4, 12, 24, 36, 52 weeks
Changes of serum IgG4 levels | At 4, 12, 24, 36, 52 weeks
security | At 4, 12, 24, 36, 52 weeks
  Use CTCAE V5.0 to record adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing 100050, Beijing, China